CLINICAL TRIAL: NCT01785758
Title: Efficacy and Safety of Sugammadex (Bridion™) in the Reversal of Profound Rocuronium-induced Neuromuscular Blockade in Patients With End-stage Renal Failure: Comparison With Healthy Patients
Brief Title: Efficacy and Safety of Sugammadex in Renal Diseased Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Hospital General Universitario Santa Lucía (Other)
Responsible Party: Principal Investigator, Camila Machado de Souza, MD, Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sugamadex01; CEP 1277/11 (Other: Federal University of Sao Paulo - Ethics Committee)
Record Dates: First submitted 2013-02-03; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Failure, Chronic; Neuromuscular Blockade
Keywords: complications, renal;; kidney, failure;; neuromuscular block, antagonism;; neuromuscular block, rocuronium;; safety, drug; sugammadex
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency | interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal Group (Experimental): Sugammadex (4mg/Kg) single dose to reverse profound neuromuscular blockade
  Interventions: Drug: Sugammadex (4 mg/Kg)
- Control group (Active Comparator): Sugammadex (4mg/Kg) single dose to reverse profound neuromuscular blockade
  Interventions: Drug: Sugammadex (4 mg/Kg)

INTERVENTIONS:
Drug: Sugammadex (4 mg/Kg) — Sugammadex administered at the end of surgical procedure, once skin suture had been finished, to reverse profound neuromuscular blockade induced and maintained with rocuronium
  Other Names: Bridion

SUMMARY:
The purpose of this study is to determine whether sugammadex reverses a profound neuromuscular blockade induced by rocuronium in patients with end-stage renal disease just as effectively and safely as it does in patients with normal renal function.

DETAILED DESCRIPTION:
Sugammadex antagonizes rocuronium induced neuromuscular blockade by encapsulating the molecules of this agent in the plasma and originating a complex which is highly stable, and mainly eliminated by the kidneys. In patients with end stage renal disease, this complex remains in the circulation for days. Previous studies have shown that sugammadex adequately reverses the blockade induced by rocuronium in such patients, and no evidence of recurrence was observed after a dosis of 2 mg/Kg administered to reverse a moderate level of blockade. To our knowledge, nothing has been published so far on the reversal of profound blockade by sugammadex in patients with renal failure.

The aim of our study was to evaluate the efficacy and safety of sugammadex in the reversal of profound neuromuscular block (NMB) induced by rocuronium in patients with end-stage renal failure and compare it to patients with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years old
* end-stage renal disease defined by clearance of creatinine < 30 ml/min
* normal renal function defined by clearance if creatinine > 90 ml/min
* candidates to elective surgical procedures (control group) or kidney transplantation (renal group) under general anaesthesia

Exclusion Criteria:

* pregnant and breastfeeding women
* patients with known or suspected neuromuscular disorders
* patients with hepatic disfunction
* a history of malignant hyperthermia
* allergy to narcotics, rocuronium or other medication used during general anaesthesia
* patients receiving medication known to interfere with the action of rocuronium (amino glycoside antibiotics, anticonvulsants, or magnesium)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Time from administration of sugammadex to recovery of the train-of-four ratio (TOF) to 0.9 | 2 hours

SECONDARY OUTCOMES:
Time from administration of sugammadex to recovery of the train-of-four ratio (TOF) to 0.7 and 0.8 | 2 hours

OTHER OUTCOMES:
Reoccurrence of neuromuscular blockade | 24 hours
  Patients will be monitored for evidence of reoccurrence of neuromuscular blockade for the first two hours after administration of sugammadex and clinically reevaluated after 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Camila M Souza, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Hospital do Rim e Hipertensão - Fundação Oswaldo Ramos, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Staals LM, Snoeck MM, Driessen JJ, Flockton EA, Heeringa M, Hunter JM. Multicentre, parallel-group, comparative trial evaluating the efficacy and safety of sugammadex in patients with end-stage renal failure or normal renal function. Br J Anaesth. 2008 Oct;101(4):492-7. doi: 10.1093/bja/aen216. Epub 2008 Jul 23. PMID 18653492
- [Background] Staals LM, Snoeck MM, Driessen JJ, van Hamersvelt HW, Flockton EA, van den Heuvel MW, Hunter JM. Reduced clearance of rocuronium and sugammadex in patients with severe to end-stage renal failure: a pharmacokinetic study. Br J Anaesth. 2010 Jan;104(1):31-9. doi: 10.1093/bja/aep340. PMID 20007792
- [Derived] de Souza CM, Tardelli MA, Tedesco H, Garcia NN, Caparros MP, Alvarez-Gomez JA, de Oliveira Junior IS. Efficacy and safety of sugammadex in the reversal of deep neuromuscular blockade induced by rocuronium in patients with end-stage renal disease: A comparative prospective clinical trial. Eur J Anaesthesiol. 2015 Oct;32(10):681-6. doi: 10.1097/EJA.0000000000000312. PMID 26225497